CLINICAL TRIAL: NCT01658800
Title: Phase I Study of the Safety and Immunogenicity of a Novel H5N1 Influenza Vaccine in Healthy Adults Age 18-49
Brief Title: Study of the Safety and Immunogenicity of a Novel H5N1 Influenza Vaccine in Healthy Adults Age 18-49
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VaxInnate Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: VAX161-01C
Record Dates: First submitted 2012-07-30; First posted 2012-08-07 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Influenza
Keywords: H5N1 Influenza; H5N1 Influenza vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- VAX161C vaccine (Experimental): Subjects will be injected into the arm on 2 occasions during the study, once on Day 0 and then again on Day 21 with the vaccine VAX161C
  Interventions: Biological: VAX161C vaccine

INTERVENTIONS:
Biological: VAX161C vaccine — Recombinant H5 influenza vaccine, VAX161C

SUMMARY:
The purpose of this study is to test an investigational vaccine known as "VAX161C." An "investigational" vaccine is one that is not licensed for commercial use in the by the United States (US) by the US Food and Drug Administration (FDA). VAX161C is a vaccine for the influenza A virus subtype H5N1 avian influenza virus (bird flu). In this study, the subject will receive the VAX161C vaccine at one of six doses to see which dose is the best. VaxInnate wants to find out how safe these doses of vaccines are and how well they are tolerated by people who receive them. To measure how effective each type of the vaccine is, VaxInnate will test the ability of the body to develop an immune response, which means how the body recognizes and defends itself against the influenza virus.

DETAILED DESCRIPTION:
SAFETY ASSESSMENTS AND REPORTING Immediate Complaints Immediate complaints are vaccination symptoms that are solicited and observed for two hours (+30 minutes) after vaccination on Day 0 and vaccination on Day 21. Solicited immediate complaints will be grouped as local (injection site) complaints and general complaints (Appendix A: Solicited Local and General Vaccination Reactogenicity Symptoms). Solicited local (injection site) complaints include redness (erythema), swelling or induration, pain, bruising and solicited general complaints will include fever, headache, fatigue, joint pain, muscle aches, shivering (chills), and increased sweating. Each of these local and general complaints will be graded for severity using the guidelines provided in Appendix B: Local Reactogenicity Toxicity Grading Scale and Appendix C: General Reactogenicity Toxicity Grading Scale. The data will be reported as "immediate complaints" and presumed to be related to the investigational product. These findings should NOT be additionally recorded as AEs unless they meet the criteria set forth in Section 8.3. Any other symptom offered by study subjects at 2 hours (+30 minutes) after each vaccination will be recorded under the AE section of the CRF.

Vaccine Reactogenicity The same sets of local and general complaints, complaints reasonably anticipated to occur as a result of receipt of the investigational product are included in the Reactogenicity Memory Aid and listed in Appendix A: Solicited Local and General Vaccination Reactogenicity Symptoms. These will be solicited by study staff in conjunction with review of the Memory Aid during the 7 days following vaccinations on Day 0 and 21. The severity will be graded using the grading scales provided in Appendix B: Local Reactogenicity Toxicity Grading Scale and Appendix C: General Reactogenicity Toxicity Grading Scale and all findings recorded in the CRFs. Symptoms from the Reactogenicity Memory Aid will be reported as "reactogenicity" and presumed to be related to the investigational product. These complaints should NOT be additionally recorded as AEs unless they meet the criteria set forth in Section 8.3. Definitions used to grade reactogenicity severity will be included on the Reactogenicity Memory Aid form.

Safety Oversight VaxInnate VaxInnate is the study Sponsor. Sponsor responsibilities will include the creation and oversight of protocol development, submission of the Investigational New Drug (IND) application to the FDA, monitoring and ensuring Good Clinical Practice (GCP) conduct of the study, and the submission of annual and final study reports to the FDA.

Safety Monitoring Committee (SMC) The SMC will consist of 3 independent medical monitors not associated with study. The Principal Investigator(s), VaxInnate Medical Monitor, and the Data Manager will provide information to the SMC. The SMC will assess the safety information after each part of the study to determine if it is safe to escalate to the next dose level. The SMC meetings will be convened after the safety data for both doses has been collected for subjects enrolled in part 1 and later for part 2. The SMC will review the safety data and make a recommendation on continuing on to the next part of the study. The safety data and the SMC's recommendations will be forwarded to CBER for their review and agreement. The SMC will also meet on an ad hoc basis to review adverse events or other safety related issues. If a safety issue occurs that would halt the study (Section 4.5), the IRB and FDA will be notified.

ANALYTICAL AND STATISTICAL ANALYSIS PLAN Data Entry and Management Subject screening/enrollment will be documented using an electronic master subject log. This log will capture the following information: subject number; initials; date screen/enroll; and, reason for not enrolling.

In this study and in VAX161B, CRFs utilizing Smart Pen TM, a digital pen technology, will be used to gather originally-captured data. Therefore, the CRFs will serve as the source documentation for all protocol procedures and assessments, except for concomitant medications, adverse events, and all "Symptom Assessments" obtained from subject-completed memory aids (MEMA CRF). For these required procedures and assessments, the collected data will be recorded onto logs or memory aids as source documentation. This data will then be transcribed onto the CRF by the study staff. Health Decisions' electronic data management system will be used to create, modify, maintain, archive, retrieve, and transmit study data.

The Investigator remains responsible for the accuracy and adequacy of all data entered onto the CRFs. Data will be monitored as described in section 10.1. Under direction of the clinical monitor, CRFs will be source document verified, as appropriate and further processed. Upon further data processing, queries may be generated and sent to the Investigator for clarification or correction. The Investigator will address any queries and resolutions verified by the clinical monitor.

The database will be "soft-locked" for analysis when all subjects' data have been entered and data queries have been resolved through Day 42 (± 2) and after immunogenicity samples have been tested.

Data Analysis Additional details of the analysis will be provided in the Statistical Analysis Plan (SAP) and the Clinical Study Report (CSR). This plan will include details of handling missing data, and if applicable, unused and spurious data. Deviations from the SAP will be reported in the CSR. The SAP will be finalized before study completion. If there are any discrepancies between the protocol and the SAP, the SAP will take precedence.

Sample Size and Power For the purpose of assessing the safety and immunogenicity of VAX161C vaccine a total of 250 subjects are divided into 6 dose groups in a ratio of 1:2:2:2:2:1. Groups of 50 subjects were chosen for the 2.5, 4, 6 and 8 µg doses, the anticipated safe and immunogenic dose range for VAX161C. Groups of 25 subjects were chosen for the 1 and 12 µg dose groups. Based on previous findings with similar vaccines, we anticipate that the 1 µg group will serve as the "placebo" group. The purpose of the 12 µg group is to assess the upper limit of safety and immunogenicity. The sample size for this study (50 subjects in each of the key vaccine doses and 25 subjects in the control (1 µg group) was selected to provide a robust initial safety database as well as some information on the dose-related immune response.

Safety Analysis All subjects who receive at least one dose of vaccine will be considered enrolled and included in the post-dosing safety analysis (safety population). The safety outcome will be the occurrence of solicited complaints (identified in Section 8.2) during the seven days after receiving the vaccine. These symptoms will be collected from the memory aid and from the information collected at the clinic visits. All symptoms will be graded according to severity. Response to vaccine will be categorized as local (arm pain, redness, bruising, etc.) or systemic (headache, muscle aches, fatigue, etc.) symptoms. Local or systemic reactions between vaccine dose groups will be compared to the 1 µg group by two-sided Fisher's exact test. Laboratory tests such as WBC and LFTs collected before and after vaccination will also be analyzed looking for differences between pre- and post-vaccination and across vaccine formats. We will compare the types and severity of symptoms and laboratory results based on vaccine construct.

Proportions for those reporting the endpoints in the vaccine groups will be calculated and analyzed using the upper boundary of a two-tailed 95% confidence interval (CI) to compare against the 1 µg group. In addition, the frequency and percent of subjects in each of the vaccine groups reporting each of the solicited complaints and laboratory findings will be tabulated and presented with 2-sided 95% confidence intervals. A chi-square test may be used to test whether the observed proportions differ from the expected proportions across dosage groups.

Immune Response Analysis

Sera collected at Screening, Days 21 (prior to vaccination0, 42 (±2) and 180 (±10) will be analyzed for determination of HAI, MN assay, serum anti-HA ELISA and serum anti-flagellin ELISA. The results of these determinations will be evaluated as follows:

* Calculation of the geometric mean of pre- and post-vaccination HAI, MN assay, anti-HA, and anti-flagellin serum antibody titers for each treatment group.
* Change from pre- to post-vaccination in geometric mean HAI, MN anti-HA, and anti-flagellin serum antibody titers for each treatment group
* Seroconversion rates based on HAI response defined as percentage of subjects having a pre-vaccination titer of < 1:10 and a post vaccination HI titer ≥ 1:40 or a pre-vaccination HI titer ≥ 1:10 and a minimum four-fold rise in post-vaccination HI antibody titer).
* Proportion of subjects with HAI, MN, anti-HA and anti-flagellin serum antibody titers before and after vaccination by treatment group.

Statistical comparisons between the treatment groups will be provided. GMTs will be compared with one-way ANOVA of log10-transformed titers and reported as GMT ratios and 95% CIs, calculated on the log10 scale and transformed. Proportions of subjects that achieve seroconversion for each dose will be determined by two-sided Fisher's exact test. Exact CIs are reported for all proportional endpoints.

Efficacy Analysis The current protocol is not designed to evaluate the efficacy of VAX161C. CLINICAL MONITORING AND ADMINISTRATION Disposition of Data A CRF will be provided for each enrolled study subject. Data collected through the completion of experimental procedures required by this protocol will be recorded in the subject's chart as source documentation. This data will then be transcribed onto the CRF by the study staff. All data entered into the CRFs will have source documentation in the form of laboratory print outs or entries into the subject's chart. The Investigator remains responsible for the accuracy and adequacy of all data entered on the CRFs. Under direction of the clinical monitor, CRFs will be source data verified and further processed. Upon further data processing, queries may be generated and sent to the Investigator for clarification or correction. The Investigator will address any queries and resolutions verified by the clinical monitor. Once all CRFs are completed and queries resolved, the subjects' CRFs may be locked.

ELIGIBILITY:
INCLUSION

* Male or female aged 18 - 49 years
* Give written informed consent
* Healthy, as determined by medical history, physical examination, vital signs, and clinical safety laboratory examinations
* Females should not be pregnant and not lactating and fulfill one of the following criteria: At least one year post-menopausal;Surgically sterile;Will use oral, implantable, transdermal or injectable contraceptives for 30 days prior to first vaccination and until 28 days after vaccination
* Willing to use another reliable form of contraception approved by the Investigator for study duration and until 28 days after vaccination.
* Women of childbearing potential must have a negative urine pregnancy test within 24 hours preceding receipt of vaccination
* Comprehension of the study requirements, expressed availability for the required study period, and ability to attend scheduled visits
* Willing to receive the unlicensed (VAX161) vaccine given as an i.m. injection.
* Willing to provide multiple blood specimens collected by venipuncture.

EXCLUSION

* Persons who have a psychiatric illness, a chronic illness, or who are taking a concomitant therapy or have any other condition that would interfere with the subject's participation in the study or interpretation of the study results.
* Persons with clinically significant abnormal liver function tests at screening.
* Positive serology for HBsAg, HCV or HIV antibodies.
* Persons having cancer or have received treatment for cancer within three years (persons with a history of cancer who are disease-free without treatment for three years or more are eligible), excluding basal cell carcinoma (BCC) or squamous cell carcinoma (SCC), which are allowed unless located at the vaccination site.
* Persons with impaired immune responsiveness, including diabetes mellitus.
* Persons presently receiving or having a recent history of receiving any medication or therapeutic modality that affects the immune system such as allergy shots, immune globulin, interferon, immunomodulators, radiation therapy, cytotoxic drugs or drugs known to be frequently associated with significant major organ toxicity, or systemic corticosteroids.
* Persons who have received or plan to receive a nonstudy vaccine within 30 days prior to vaccination and during 42 day study period following vaccination, including licensed influenza vaccines.
* history of anaphylactic type reaction to injected vaccines.
* history of drug or chemical abuse in the year prior to screening.
* history of Guillain-Barré Syndrome.
* have received, or plan to receive, any investigational product or non-registered drug within 30 days prior to vaccination and during the 42 day study period after vaccination.
* Receipt of blood or blood products 8 weeks prior to vaccination or planned administration during the 42 day study period following vaccination.
* Donation of blood or blood products within 8 weeks prior to vaccination or at any time during the study.
* Acute disease within 72 hours prior to vaccination, defined as the presence of a moderate or severe illness with or without fever, or a fever > 100.4° F orally.
* significant cardiovascular disease e.g., New York Heart Association (NYHA) Class 3 or 4 congestive heart failure; myocardial infarction within the past six months; unstable angina, coronary angioplasty within the past six months; uncontrolled ventricular cardiac arrhythmias; resting heart rate (HR) >100 beats per minute (bpm).
* history of chronic obstructive pulmonary disease or history of other lung disease.
* Any condition that, in the opinion of the investigator, might interfere with study objectives.
* Previously received an H5 or avian influenza vaccine, including VAX161.
* Persons with a BMI ≥40

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 275 (Actual)
Dates: Start 2012-09; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Safety | 1 year
  Assess safety, reactogenicity and tolerability. Symptoms will be collected from the memory aid adn from the information collected at the clinic visits. All symptoms will be graded according to severity. Response to vaccine will be categorized as local (arm pain, redness, bruising, etc.) or systemic (headace, muscle aches, fatigue, etc.) symptoms. Laboratory tests such as CRP, WBC, LFTs and cytokines collected before and after vaccination will also be analyzed. We will compare the types and severity of symptoms and laboratory results based on vaccine dose.

SECONDARY OUTCOMES:
Immunogenicity | 6 months
  To assess serum immune response, sera collected at Days 0, 21, 42 and 180 will be analyzed for HAI, MN, serum IgG anti-HA and serum IgG anti-flagellin by Elisa. The geometric mean, seroconversion and seroprotection rates will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: David Taylor, MD, Study Director — VaxInnate Corporation
Locations (2):
- United States (2):
  - Miami Research Associates, South Miami, Florida
  - Johnson County Clinical Trials, Lenexa, Kansas